CLINICAL TRIAL: NCT04351022
Title: Pilot Study of the Efficacy and Safety of CD38 Targeted Chimeric Antigen Receptor Engineered T-Cells in the Treatment of CD38 Positive Relapsed or Refractory Acute Myeloid Leukemia (AML)
Brief Title: CD38-targeted Chimeric Antigen Receptor T Cell (CART) in Relapesd or Refractory Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UnicarTherapy2020001
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: CD38, CART, AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD38 positive relapsed or refractory acute myeloid leukemia (Experimental)
  Interventions: Biological: CART-38

INTERVENTIONS:
Biological: CART-38 — Split intravenous infusion of CART-38 cells [dose escalating infusion of (5-20)x10^6 CART-38 cells/kg].

SUMMARY:
This is a single center, open-label phase 1/2 study to evaluate the safety and efficacy of targeted CD38 chimeric antigen receptor engineered T cell immunotherapy (CART) in the treatment of CD38 positive relapsed or refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
The patients will receive infusion of CAR T-cells targeting CD38 to confirm the safety and efficacy of CD38 CAR T-Cells in relapsed or refractory acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

* CD38 positive relapsed/refractory acute myeloid leukemia
* age 6-65 years.
* left ventricular ejection fractions ≥ 0.5 by echocardiography
* creatinine < 1.6 mg/dL
* aspartate aminotransferase/aspartate aminotransferase < 3x upper limit of normal
* Total bilirubin <2.0 mg/dL
* karnofsky performance status ≥ 60
* expected survival time ≥ 3 months (according to investigator's judgement)

Exclusion Criteria:

* patients are pregnant or lactating
* uncontrolled active infection
* class III/IV cardiovascular disability according to the New York Heart Association Classification
* active hepatitis B or hepatitis C infection
* patients with HIV infection
* patients with history of seizure
* active central nervous system leukemia

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events | 12 months
  Adverse events are evaluated with CTCAE V5.0

SECONDARY OUTCOMES:
Overall response rate (ORR) | 2 years
  ORR includes CR, CRi, MLFS and PR. Complete remission (CR)：Bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count >1.0x 10^9/L; platelet count >100x10^9/L. CR with incomplete hematologic recovery (CRi)：All CR criteria except for residual neutropenia (<1.0x10^9/L) or thrombocytopenia (<100x10^9/L). Morphologic leukemia-free state (MLFS): Bone marrow blasts <5%; absence of blasts with Auer rods; absence of extramedullary disease; no hematologic recovery required. Partial remission (PR): All hematologic criteria of CR; decrease of bone marrow blast percentage to 5% to 25%; and decrease of pretreatment bone marrow blast percentage by at least 50%.
Event-free survival (EFS) | 2 years
  time from enrollment to the date of primary refractory disease, or relapse from CR or CRi, or death from any cause.
Cumulative incidence of relapse(CIR) | 2 years
  time from the date of achievement of a remission until the date of relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowen Tang, Ph.D, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cui Q, Liang P, Dai H, Cui W, Cai M, Ding Z, Ma Q, Yin J, Li Z, Liu S, Kang L, Yao L, Cen J, Shen H, Zhu M, Yu L, Wu D, Tang X. Case report: CD38-directed CAR-T cell therapy: A novel immunotherapy targeting CD38- positive blasts overcomes TKI and chemotherapy resistance of myeloid chronic myeloid leukemia in blastic phase. Front Immunol. 2022 Nov 29;13:1012981. doi: 10.3389/fimmu.2022.1012981. eCollection 2022. PMID 36524116
- [Derived] Cui Q, Qian C, Xu N, Kang L, Dai H, Cui W, Song B, Yin J, Li Z, Zhu X, Qu C, Liu T, Shen W, Zhu M, Yu L, Wu D, Tang X. CD38-directed CAR-T cell therapy: a novel immunotherapy strategy for relapsed acute myeloid leukemia after allogeneic hematopoietic stem cell transplantation. J Hematol Oncol. 2021 May 25;14(1):82. doi: 10.1186/s13045-021-01092-4. PMID 34034795